CLINICAL TRIAL: NCT01766492
Title: Quality of Life in Patients With Clinically Localized Prostate Cancer Treated With Stereotactic Body Radiation Therapy (SBRT)
Brief Title: Quality of Life in Patients With Clinically Localized Prostate Cancer Treated With Radiosurgery
Acronym: PR-PROS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-1175
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer; Localized Malignant Neoplasm
Keywords: prostate cancer; CyberKnife
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- male (age > 18 y/o) with prostate cancer: Men received Stereotactic Body Radiation Therapy (SBRT) for clinically localized prostate cancer
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic body radiation therapy for prostate
  Other Names: CyberKnife radiosurgery

SUMMARY:
Quality of life data following SBRT for prostate cancer has been obtained in only a small numbers of patients. A prospective study using validated quality of life questionnaires is needed to determine outcomes after treatment with SBRT. Our study will be the first essential step in developing a better evidence base on the comparative risks and benefits of SBRT treatment with regards to quality of life assessment and outcomes.

DETAILED DESCRIPTION:
Study Design (for example, hypothesis, research question, standard and experimental procedures, special or unusual equipment or procedures):

The main goal of this study is to evaluate quality of life outcomes and changes in patient reported symptoms (e.g. urinary, bowel and sexual function) in patients receiving SBRT treatment for clinically localized prostate cancer. Validated quality of life questionnaires will be administered in a deidentified, prospective fashion. Eligible subjects will be patients undergoing SBRT treatment for prostate cancer.

Hypothesis: Patients undergoing SBRT will have similar cancer control and symptoms as men who are treated with other radiation therapy modalities.

Primary objective: To evaluate quality of life outcomes (e.g. fatigue, urinary, bowel and sexual function) for patients with clinically localized prostate cancer treated with SBRT.

Secondary objectives: Prospective data on cancer control and toxicity following SBRT for clinically localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of prostate
* Signed study-specific consent
* Prostate Specific Antigen (PSA) within 60 days of registration

Exclusion Criteria:

* Prior pelvic radiotherapy
* Prior radical prostate surgery
* Medical or psychiatric illness that would interfere with treatment or follow up
* Implanted hardware adjacent to the prostate that would prohibit appropriate treatment planning and/or treatment delivery

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men (> 18 y/o) with clinically localized prostate cancer,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
fatigue | 2 years
  Use questionnaire to assess patient's symptoms regarding fatigue
urinary symptoms | 24 months
  Use questionnaire to assess patient's symptoms regarding urinary symptoms after radiosurgery
bowel symptoms | 24 months
  Use questionnaire to assess patient's symptoms regarding bowel symptoms after radiosurgery
sexual function | 24 months
  Use questionnaire to assess patient's symptoms regarding sexual symptoms after radiosurgery

SECONDARY OUTCOMES:
cancer control | 24 months
  clinical evidence of localized and distal cancer controls
toxicity symptoms | 24 months
  Evaluate all the treatment-related toxicity by both clinical evidence(physical exam and lab) and quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Collins, MD, PhD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
NO individual data will be made available

REFERENCES:
- [Background] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880
- [Derived] Dess RT, Devasia TP, Aghdam N, Jackson WC, Soni PD, Smith CP, Mitchell AL, Suy S, Hamstra DA, Jolly S, Nguyen PL, Feng FY, Schipper MJ, Skolarus TA, Miller DC, Wittmann DA, Collins SP, Spratt DE. Patient-Reported Sexual Aid Utilization and Efficacy After Radiation Therapy for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2018 Jun 1;101(2):376-386. doi: 10.1016/j.ijrobp.2018.01.055. Epub 2018 Jan 31. PMID 29487023